CLINICAL TRIAL: NCT04670770
Title: An Open Label Phase II Clinical Trial Evaluating the Efficacy and Safety of SHR1459 in Adult Patients With Neuromyelitis Optical Spectrum Disorders (NMOSDs)
Brief Title: An Open Label Study of the Effects of SHR1459 in NMOSDs Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSB20621
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR1459 (Experimental): SHR1459
  Interventions: Drug: Drug - SHR1459

INTERVENTIONS:
Drug: Drug - SHR1459 — Oral Tablets taken once daily for 52 weeks

SUMMARY:
This is an open-label study, to evaluate the efficacy and safety of SHR1459 in participants with NMOSDs.

DETAILED DESCRIPTION:
Therefore, the investigators of this study are investigating whether SHR1459 could prevent relapse of NMOSDs.

The primary objective of this study is to evaluate the effectiveness of SHR1459 in NMOSDs patients.

The secondary objectives are to determine:

The safety profile of SHR 1459 in patients with NMOSDs. Whether SHR1459 reduce MRI lesions and APQ4-Abs level.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age.
2. Diagnosis of AQP4-IgG positive NMOSD according to IPND diagnostic criteria 2015 at screening.
3. Having a documented history of 2 or more NMOSD relapse required rescue therapy(ies) within the last 12 months.
4. Subjects must be stable treatment (if any) for more than 1 month before starting the IP treatment, which is defined as follows:- Expanded disability status scale (EDSS) score≦7.5
5. Written informed consent obtained before any study procedure.
6. Subjects are willing and able to comply with the visit schedule and treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Allergic to the investigative product or any ingredient in the investigative product.
2. Past or current malignancy, except for cutaneous non-metastatic basal cell carcinoma or squamous cell carcinoma that has been adequately treated or removed
3. The subject currently has a central nervous system (CNS) disease that may affect the assessment of NMOSD;
4. Severe and uncontrolled conditions that the investigator determines may affect subjects' safety, trial compliance, evaluation of the end point, or the need to use medications not permitted in the protocol;
5. The investigator judges that the subject has a disease that affects the absorption, distribution, metabolism and excretion of the drug;
6. The subjects had any major clinical infection and was hospitalized or treated with parenteral antibiotics within 1 month before screening; Or other infections that investigator thought might aggravate as a result of participating in the study;
7. The subject may have an active, latent or undertreated Mycobacterium tuberculosis (ie, tuberculosis [TB]) infection, defined as follows:

   * The result of QuantiFERON-TB Gold (QFT Gold test) was positive or the result of T-SPOT.TB was positive within 3 months before screening/screening period.
   * Or chest imaging examinations suggest the presence of active tuberculosis infection within 3 months before screening / during the screening period;
   * The result of QuantiFERON-TB Gold (QFT Gold test) was positive or the result of T-SPOT.TB was positive within 3 months before screening/screening period.
   * Or chest imaging examinations suggest the presence of active tuberculosis infection within 3 months before screening / during the screening period;
8. Positive laboratory tests related to human immunodeficiency virus (HIV) or hepatitis B virus or hepatitis C virus;
9. Have received BTK inhibitors (e.g. ibrutinib) at any time in the past.
10. Received B-cell targeted therapy (such as rituximab) within 12 weeks before the first administration.
11. Received biological agents such as eculizumab, tocilizumab, Satralizumab, Alemtuzumab, Natalizumab within 12 weeks before the first administration;
12. Subjects who may receive any live attenuated vaccine during the screening period or have received any live virus vaccine within 8 weeks prior to initial administration;
13. Any concomitant disease other than NMOSD that requires glucocorticoid therapy (oral or IV) within the 6 months prior to screening.
14. Abnormal and clinically significant ECG examination during screening.
15. Alanine glutamate aminotransferase (ALT)>2 times the upper limit of normal (ULN) and/or glutamate aspartate aminotransferase (AST)>2 times ULN and/or bilirubin>2 times ULN during the screening period ULN;
16. Abnormal white blood cell count, neutrophil count, lymphocyte count, or platelet count during the screening period are considered unsuitable for participating in the study after the investigator's assessment (refer to the following criteria):

    * Hemoglobin <100 g/L or hematocrit <30%;
    * White blood cell (WBC) count<3.0×109/L (<3000/mm3) or ANC<1.2×109/L (<1200/mm3);
    * Lymphocytes <0.8×109/L (<800/mm3);
    * Platelet count<100×109/L (<100,000/mm3)
17. eGFR≤60 ml/min (calculated according to Cockcroft-Gault) or receiving dialysis during the screening period.
18. Unable to undergo MRI scans. History of clinically significant CNS trauma (e.g. traumatic brain injury, cerebral contusion, spinal cord compression)
19. Pregnant or breastfeeding women;
20. Use of an investigational drug or other experimental therapy within 4 weeks, 5 pharmacokinetic half-lives, or the duration of biological effect (whichever is longer) prior to screening.
21. Any other conditions in which the investigator or sponsor believes that the subject is not suitable for inclusion in the study.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of SHR1459 in patients with relapsing NMOSDs | 52 weeks
  Comparison of the annualized relapse rate at 52 weeks of treatment with the annualized recurrence rate before screening.

SECONDARY OUTCOMES:
Comparison of the annualized relapse rate at 52 weeks of treatment with the year before screening. | 52 weeks
  Comparison of the annualized relapse rate at 52 weeks of treatment with the year before screening.
Proportion of subjects who are relapse-free at week 24 and 52. | 52 weeks
  Proportion of subjects who are relapse-free at week 24 and 52.
Changes in the expanded disability status scale (EDSS) at week 4, 12, 24, 36, and 52 compared to baseline. | 52 weeks
  Changes in the expanded disability status scale (EDSS) at week 4, 12, 24, 36, and 52 compared to baseline.
Changes in low-contrast visual acuity (LCVA) score at week 4, 12, 24, 36 and 52 compared to baseline | 52 weeks
  Changes in low-contrast visual acuity (LCVA) score at week 4, 12, 24, 36 and 52 compared to baseline.
Changes in cumulative active MRI lesion count at week 24 and 52 compared to baseline. | 52 weeks
  Changes in cumulative active MRI lesion count at week 24 and 52 compared to baseline.
Changes in health related quality of life (HRQoL) at week 12, 24, 36 and 52 compared to baseline. | 52 weeks
  Changes in health related quality of life (HRQoL) at week 12, 24, 36 and 52 compared to baseline.
Changes in pain severity score (NRS) at week 4, 12, 24, 36 and 52 compared to baseline. | 52 weeks
  Changes in pain severity score (NRS) at week 4, 12, 24, 36 and 52 compared to baseline.
Changes in serum AQP4-IgG titer from baseline at 4, 12, 24, 36, 52 weeks. | 52 weeks
  Changes in serum AQP4-IgG titer from baseline at 4, 12, 24, 36, 52 weeks.
Changes in the absolute value of B lymphocytes and total immunoglobulins (IgA, IgG and IgM) from baseline after 12, 24, and 52 weeks of treatment. | 52 weeks
  Changes in the absolute value of B lymphocytes and total immunoglobulins (IgA, IgG and IgM) from baseline after 12, 24, and 52 weeks of treatment
The plasma concentration of SHR1459 and its metabolite SHR1459-02 in NMOSD patients. | 52 weeks
  The plasma concentration of SHR1459 and its metabolite SHR1459-02 in NMOSD patients

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Xiangya Hospital Of Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Lanzhou University Second Hospital, Lanzhou
  - People's Hospital of Rizhao, Rizhao
  - Huashan Hospital Affiliated To Fudan University, Shanghai
  - First Hospital Of Shanxi Medical University, Taiyuan
  - Tangdu Hosiptal, Xi'an
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No